CLINICAL TRIAL: NCT05642806
Title: Comparison of Immune Profiles in Chronic Rhinosinusitis Patients After Mepolizumab Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Paul's Sinus Centre (Other)
Responsible Party: Principal Investigator, Dr. Andrew Thamboo, MD, Clinical Assistant Professor, St. Paul's Sinus Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H20-03358
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Asthma; Chronic Rhinosinusitis Without Nasal Polyps
Keywords: asthma; chronic rhinosinusitis; nasal polyps; mepolizumab
MeSH Terms: conditions — Asthma; Nasal Polyps | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study pharmacist and one of the research coordinators will be unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepolizumab (Experimental): Mepolizumab (100 mg) subcutaneously every 4 weeks
  Interventions: Biological: Mepolizumab
- Placebo (Placebo Comparator): Placebo 100 mg subcutaneously every 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab will be administered subcutaneously (SC) every 4 weeks for a total of 24 weeks
  Arms: Mepolizumab
Other: Placebo — Placebo will be administered subcutaneously (SC) every 4 weeks for a total of 24 weeks
  Arms: Placebo

SUMMARY:
This study aims to analyze the immune profiles of patients with Chronic Rhinosinusitis with Nasal polyps (CRSwNP) with and without asthma before and after Mepolizumab.

A group of participants with CRS without nasal polyps (CRSsNP) with asthma will be included to compare their immune profiles to CRSwNP.

DETAILED DESCRIPTION:
The proposed design is a 24-week randomized, double-blind, placebo-controlled, parallel-group study to compare the molecular profiles of CRSwNP patients with or without asthma after Mepolizumab treatment. Subjects must sign an informed consent before any study-related procedure is performed. At visit 1 (Screening) nasoendoscopy procedure, blood test analysis, and asthma history evaluation will be performed for all subjects. Newly diagnosed asthma patients will be confirmed by specific tests (methacholine and atopy test) between screening and baseline visits. Subjects who meet eligibility criteria at Visit 2 (Baseline) will be randomized to receive either mepolizumab or placebo in addition to standard-of-care CRS treatment using block randomization through REDCap. This study will be blinded to the PI, the patient, and one of the research coordinators. The blinded research coordinator will be responsible for randomizing the study subjects using REDCap.

In this visit, a nasal sample will be collected to measure the analysis of the inflammatory cytokine from the nasal secretions. This procedure will be repeated in the middle and end of treatment (week 8 and week 24). During the blind-treatment run-in period, study treatment will be administered at St Paul's Hospital every 4 weeks for 6 months. Participants will complete different questionnaires to measure the symptoms and social/emotional consequences of the subject's nasal disorder (SNOT- 22), health-related quality of life EuroQol-5 (EQ-5D), and an objective smell identification test (SIT). They will assess their global impression of change since starting the study drug using the Patient Global Impression of Change (PGIC) scale.

This study will also include 30 participants with CRSsNP with asthma that will not undergo any study procedure except the Screening and Baseline Visit to collect a nasal sample for cytokine analysis. These results will later be compared to those who positively responded to Mepolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Are over the age of 19.
2. Patients with CRSwNP with or without asthma:

   * Asthma confirmed with a spirometry and assessment on previous history of asthma (a methacholine challenge test and atopy testing to document positive or negative history of asthma will be performed if there is no clinical record).
   * Presence or absence of nasal polyps. This can be based on formal exam at Baseline Visit or historical assessment.
3. Patients with CRSsNP with asthma:

   * These patients will not take the study treatment and they will only complete screening and baseline visits.
4. Females of childbearing potential must commit to using an acceptable method of birth control for the duration of the study and they must have a negative urine pregnancy test at each study visit.

Exclusion Criteria:

1. Current or past sinonasal or bronchial tumours
2. Subjects who have been treated with oral antibiotics in the past month prior to surgery.
3. Subjects with known immunodeficiency
4. Subjects with known autoimmune disease
5. Smoking history; current or former smokers.
6. Prior lung transplants
7. Subjects with parasitic (helmintic) infection
8. Subjects with hypersensitivity; with allergy/intolerance to a monoclonal antibody or biologic
9. Female participants who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the immune profile in CRSwNP patients with and without asthma (before and after Mepolizumab treatment), and with asthmatic CRSsNP patients. | 24 weeks
  • Mean change from baseline in key inflammatory cytokines measured by the Luminex Bio-Plex Pro Human Cytokine Multi-Plex (the specific cytokine targets for this assay include: IL-1β, IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17, basic FGF, eotaxin, G-CSF, GM-CSF, IFNγ, IP-10, MCP-1 (MCAF), MIP-1α, MIP-1β, PDGF-BB, RANTES, TNF-α, VEGF)

SECONDARY OUTCOMES:
Explore the effects of Mepolizumab compared to placebo in the treatment of Chronic Rhinosinusitis | 24 weeks
  Mean change from baseline in Modified Lund-Kennedy (MLK) endoscopic scores
Explore the effects of Mepolizumab compared to placebo in the treatment of Chronic Rhinosinusitis | 24 weeks
  Mean change from baseline in the 22-item Sino Nasal Outcome Test (SNOT-22)
Examine the treatment response to Mepolizumab in CRSwNP patients with and without asthma. | 24 weeks
  Mean change from baseline in MLK
Examine the treatment response to Mepolizumab in CRSwNP patients with and without asthma. | 24 weeks
  Mean change from baseline in SNOT-22

CONTACTS AND LOCATIONS:
Locations (1):
- St. Pual's Sinus Centre, Vancouver, British Columbia, Canada